CLINICAL TRIAL: NCT02041273
Title: A Phase 1, Open-label 6 Sequence 3 Period Crossover Study of Palbociclib (PD- 0332991) in Healthy Volunteers to Estimate the Relative Bioavailability of Palbociclib Formulations
Brief Title: Relative Bioavailability Of Palbociclib (PD-0332991) Under Fed And Fasted Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: A5481036
Record Dates: First submitted 2014-01-14; First posted 2014-01-22 (Estimated); Last update posted 2014-03-17 (Estimated); Status verified 2014-03

CONDITIONS: Healthy
Keywords: bioavailability; bioequivalence; AUC; Cmax
MeSH Terms: interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Palbociclib given to healthy volunteers (Experimental)
  Interventions: Drug: palbociclib isethionate (phase 1 and 2 studies); Drug: palbociclib commercial free base capsule

INTERVENTIONS:
Drug: palbociclib isethionate (phase 1 and 2 studies) — 125 mg palbociclib isethionate salt under overnight fasting conditions
Drug: palbociclib isethionate (phase 1 and 2 studies) — 125 mg palbociclib isethionate salt under minimal fasting conditions (1 hr before palbociclib administration and 2 hrs post dose)
Drug: palbociclib commercial free base capsule — 125 mg palbociclib commercial free base capsule under fed conditions ( moderate fat meal)

SUMMARY:
A relative bioavailability study of commercial palbociclib free base hard capsules to the isethionate salt palbociclib capsules ( used in Phase 1 and 2 studies) under different fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects and/or female subjects of non-childbearing potential between the ages of 18 and 55 years.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
* Any condition possibly affecting drug absorption.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - 8)] | 7 days
  AUC (0 - 8)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 8). It is obtained from AUC (0 - t) plus AUC (t - 8).
Maximum Observed Plasma Concentration (Cmax) | 7 days

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | 7 days
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Apparent Oral Clearance (CL/F) | 7 days
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Plasma Decay Half-Life (t1/2) | 7 days
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Apparent Volume of Distribution (Vz/F) | 7 days
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5481036&StudyName=Relative%20Bioavailability%20Of%20%20Palbociclib%20%28PD-0332991%29%20Under%20Fed%20And%20Fasted%20Conditions